CLINICAL TRIAL: NCT06347653
Title: A Single Arm, Open Label, Multicenter Clinical Trial of Linperlisib Combined With CHOP Regimen Followed by Autologous Hematopoietic Stem Cell Transplantation and Linperlisib Monotherapy Maintenance for Newly Diagnosed Nodal T-follicular Helper Cell Lymphoma (nTFHL) Patients
Brief Title: Linperlisib-based Treatment Regimen in Newly Diagnosed Nodal T-follicular Helper Cell Lymphoma (nTFHL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023KT127
Record Dates: First submitted 2023-07-13; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Nodal T-follicular Helper Cell Lymphoma
Keywords: nodal T-follicular helper cell lymphoma; linperlisib; autologous hematopoietic stem cell transplantation; maintenance treatment
MeSH Terms: interventions — VAP-cyclo protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- linperlisib combined with CHOP regimen (Experimental)
  Interventions: Drug: linperlisib combined with CHOP regimen

INTERVENTIONS:
Drug: linperlisib combined with CHOP regimen — Induction therapy: cyclophosphamide 750 mg/m2 day1, doxorubicin 40-50 mg/m2 day1, vincristine 1.4 mg/m2 (max 2 mg) day1, prednisone 100 mg day1-5, linperlisib 80mg once a day，day1-21, repeat every 21 days, for 6 cycle.
  Consolidation therapy: high dose chemotherapy followed by autologous hematopoietic stem cell transplantation.
  Maintenance therapy: linperlisib 80 mg day1-28, up to 12 cycles.

SUMMARY:
This study is conducted to evaluate the efficacy and safety of linperlisib combined with CHOP regimen followed by autologous hematopoietic stem cell transplantation and linperlisib monotherapy maintenance for newly diagnosed nTFHL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed nTFHL classified by WHO-HAEM5, including nodal TFH cell lymphoma, angioimmunoblastic-type, nodal TFH cell lymphoma, follicular-type, Nodal TFH cell lymphoma, NOS
2. Patients planning to receive autologous hematopoietic stem cell transplantation;
3. No previous systemic treatment before enrollment.;
4. There is at least one measurable lesion: the longest diameter (LDi) of the lymph node lesion is greater than 1.5 cm, or the LDi of one extra lymph node lesion is greater than 1 cm (according to the 2014 Lugano classification);
5. Age range from 18 to 65 years old, regardless of gender;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)≤2;
7. Expected survival time≥12 weeks;
8. Adequate bone marrow and organ functions; For female participants of childbearing period, a negative urine or serum pregnancy test should be performed with 1 week prior to receiving first dose of investigational drug (day 1 of cycle 1). If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required.WOCBP subjects and male subjects whose partners are WOCBP should agree to use effective contraception from the time of signing the ICF until 6 months after the last dose of study drug.
9. Adequate organ and bone marrow function without severe hematopoietic abnormalities and abnormal heart, lung, liver, kidney, thyroid function and immunodeficiencies (no blood transfusion, granulocyte colony-stimulating factor or other related medical support within 14 days prior to administration of study drug):

   1. Routine blood tests (not transfused, not on granulocyte colony-stimulating factor (G-CSF), not corrected with medication within 14 days prior to screening): hemoglobin (Hb) ≥ 90 g/L; neutrophils (ANC) ≥ 1.5 x 10 9/L; platelets (PLT) ≥ 100 x 109/L;
   2. Biochemical tests: TBIL <1.5 × upper limit of normal range (ULN); glutamate alanine aminotransferase (ALT) and glutamate aspartate aminotransferase (AST) ≤2.5 × ULN; serum creatinine (Cr) ≤1.25 × ULN or endogenous creatinine clearance ≥60 mL/min (Cockcroft-Gault formula);
   3. Coagulation (unless the subject is receiving anticoagulant therapy and coagulation parameters (PT/INR and APTT) are within the expected range for treatment with anticoagulants at screening): international normalized ratio (INR) ≤ 1.5 x ULN; activated partial thromboplastin time (APTT) ≤ 1.5 x ULN.
10. Volunteer to participate in clinical research and sign an informed consent form, willing to follow and capable of completing all trial procedures.

Exclusion Criteria:

If a patient has any of the following conditions should not be included in this study:

1. Known allergy to the active ingredients or excipients of linperlisib and CHOP regimens.
2. Patients with factors that affect oral medications (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
3. Medical History and comorbidity

   1. The subject had any active, known, or suspected autoimmune disease. Subjects who are in a stable state and do not require systemic immunosuppressive therapy are admitted;
   2. Known history of interstitial pneumonia;
   3. Current or previous history of other malignancies within 2 years prior to study enrollment.Radically treated basal cell carcinoma of the skin, papillary thyroid carcinoma, squamous skin carcinoma, carcinoma in situ of the breast and carcinoma in situ of the cervix, excepted
   4. Received systemic antitumor therapy, including chemotherapy, immunotherapy, and biotherapy (tumor vaccines, cytokines, or growth factors used to control cancer) within 28 days prior to study enrollment.
   5. Received autologous or allogeneic hematopoietic stem cell transplantation;
   6. Patients with active tuberculosis (TB) should be excluded.
   7. Severe acute or chronic infections requiring systemic treatment;
   8. Patients with hypertension that is not well controlled with antihypertensive medications (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
   9. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
   10. Patients with heart failure (New York Heart Association standard Class III or IV), poor coronary artery disease control or arrhythmia, or a history of myocardial infarction within the 6 months prior to screening despite receiving appropriate medication;
   11. Had clinically significant bleeding symptoms or definite bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, stool occult blood ++ or above at baseline, or vasculitis;
   12. Renal failure requiring hemodialysis or peritoneal dialysis;
   13. Urine routine indicated urinary protein ≥++, and 24-hour urinary protein quantity > 1.0 g；
   14. Patients who have had major surgery or severe trauma have had the effects of the surgery or trauma resolved for less than 28 days prior to enrollment；
   15. Complicated interstitial lung disease or history of severely impaired lung function;
   16. Patients requiring systemic therapy with corticosteroids (> 10 mg/day of prednisone or equivalent) or other immunosuppressive agents within 14 days prior to administration of study drug. Inhaled or topical steroids and adrenal hormone replacement at doses > 10 mg/day prednisone efficacy dose are allowed in the absence of active autoimmune disease;
4. Physical and laboratory findings

   1. A known history of human immunodeficiency virus (HIV) infection (i.e., HIV antibody positive).
   2. Active hepatitis [Hepatitis B: Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) positive and ALT above the upper limit of detection; Hepatitis C: Hepatitis C virus (HCV) ribonucleic acid (RNA) positive and ALT above the upper limit of detection]; co-infection with Hepatitis B and Hepatitis C;
5. Any medical history or disease evidence that may interfere with the study results or other conditions that investigators consider inappropriate for the study.
6. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 year
  PFS will be calculated from the start of study drug treatment to the date of disease progression, death, or last follow-up, as appropriate.

SECONDARY OUTCOMES:
ORR | After 6 cycles of induction therapy ，average of 4.2 month and post transplantation
  ORR is defined as sum of CR and PR rates, as assessed by the Investigator according to the Lugano Classification
CR rate | After 6 cycles of induction therapy ，average of 4.2 month and post transplantation
  CR rate is defined as the percentage of patients showing complete response as assessed by the Investigator according to the Lugano Classification.
Success rate of stem cell collection | 1day before performing an autologous hematopoietic stem cell transplant
  Success rate was assessed as the number of participants who achieved the target collection of CD34+cells ≥ 2×10^6/kg .
overall survival (OS) | 2 year
  OS will be calculated from the start of study drug treatment to the date of disease death or last follow-up, as appropriate.
time to next anti-lymphoma treatment | 2 year
  TTNLT will be calculated from the start of study drug treatment to the date of starting next anti-lymphoma treatment
adverse events | Toxicity will be graded according to the NCI-CTCAC version 4.0, from the first day of the first cycle of induction therapy to 30 days after the last dose of study drug.
  incidence of adverse event, proportion of patients with dose adjustment of linperlisib

CONTACTS AND LOCATIONS:
Overall Officials: PING WEI LIU, Master, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Bejing Cancer Hospital, Beijing, Beijing Municipality, China